CLINICAL TRIAL: NCT02053948
Title: Randomized Clinical Trial of Stoma Reversal Comparing Pursestring Wound Closure vs "Gunsight" Skin Incision and Closure Technique to Eliminate the Risk of Wound Infection
Brief Title: Pursestring Wound Closure vs "Gunsight" Skin Incision and Closure Technique to Reverse Stoma
Acronym: GSICT1126
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Beijing Friendship Hospital (Other); Shengjing Hospital (Other); Hebei Medical University Fourth Hospital (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Peking University People's Hospital (Other); Peking Union Medical College Hospital (Other); Chinese PLA General Hospital (Other); Jinling Hospital, China (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Zhen Jun Wang, Professor, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GSICT1126
Record Dates: First submitted 2013-11-26; First posted 2014-02-04 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Colostomy
Keywords: Reversal; Surgical technique; Pursestring Wound Closure; Gunsight Skin Incision and Closure Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pursestring Wound Closure group (Experimental): use Pursestring Wound Closure technique to close the stoma
  Interventions: Procedure: Pursestring Wound Closure
- Gunsight Skin Incision and Closure group (Experimental): use Gunsight Skin Incision and Closure Technique to close the stoma
  Interventions: Procedure: Gunsight Skin Incision and Closure Technique

INTERVENTIONS:
Procedure: Pursestring Wound Closure
  Arms: Pursestring Wound Closure group
Procedure: Gunsight Skin Incision and Closure Technique
  Arms: Gunsight Skin Incision and Closure group

SUMMARY:
The use of temporary stomas has been demonstrated to reduce septic complications after colorectal cancer surgery, especially in high-risk anastomosis; therefore, it is necessary to reduce the number of complications secondary to ostomy takedowns, namely wound infection. The aim of this study is to compare the rates of superficial wound infection, healing time and patient satisfaction after pursestring closure vs "gunsight" skin incision and closure technique closure.

ELIGIBILITY:
Inclusion Criteria:

* loop colostomy
* end colostomy

Exclusion Criteria:

* other stomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-11-30; Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
superficial wound infection of stoma site | 1 year

SECONDARY OUTCOMES:
Healing time after stoma reversal | 1 year

OTHER OUTCOMES:
Patient's satisfaction about the wound after stoma reversal | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jiagang Han, Professor, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Camacho-Mauries D, Rodriguez-Diaz JL, Salgado-Nesme N, Gonzalez QH, Vergara-Fernandez O. Randomized clinical trial of intestinal ostomy takedown comparing pursestring wound closure vs conventional closure to eliminate the risk of wound infection. Dis Colon Rectum. 2013 Feb;56(2):205-11. doi: 10.1097/DCR.0b013e31827888f6. PMID 23303149
- [Background] Lim JT, Shedda SM, Hayes IP. "Gunsight" skin incision and closure technique for stoma reversal. Dis Colon Rectum. 2010 Nov;53(11):1569-75. doi: 10.1007/DCR.0b013e3181f0535a. PMID 20940608
- [Derived] Han JG, Yao HW, Zhou JP, Zhang H, Wang GY, Shen ZL, Gong JF, Wang ZJ; Colorectal Surgery Group of Chinese Academic Society of Young Surgeons. Gunsight Procedure Versus the Purse-String Procedure for Closing Wounds After Stoma Reversal: A Multicenter Prospective Randomized Trial. Dis Colon Rectum. 2020 Oct;63(10):1411-1418. doi: 10.1097/DCR.0000000000001755. PMID 32969884
- See also: the Technique used in this trial — http://www.ncbi.nlm.nih.gov/pubmed/